CLINICAL TRIAL: NCT03809117
Title: A Randomized Controlled Trial of Biofire Film Array Gastrointestinal Panel Compared to Usual Care for Evaluation of Acute Infectious Diarrhea in the Emergency Department
Brief Title: Film Array Gastrointestinal Panel Compared to Usual Care for ED Evaluation of Infectious Diarrhea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was halted due to obstacles faced in executing clinical procedures as a result of the COVID-19 pandemic.
Sponsor: Andrew Meltzer (Other)
Collaborators: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor-Investigator, Andrew Meltzer, Associate Professor of Emergency Medicine, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #051839
Record Dates: First submitted 2018-11-13; First posted 2019-01-18 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Infectious Diarrhea
MeSH Terms: conditions — Dysentery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental (Experimental): Gastrointestinal Polymerase Chain Reaction test performed and results communicated to treatment provider. Followed by usual care per treating physician.
  Interventions: Diagnostic Test: Biofire Film Array Gastrointestinal Panel
- Control (Active Comparator): Gastrointestinal Polymerase Chain Reaction test performed at the conclusion of the study. Clinician will not be informed of results. Usual Care performed per treating physician.
  Interventions: Diagnostic Test: Biofire Film Array Gastrointestinal Panel

INTERVENTIONS:
Diagnostic Test: Biofire Film Array Gastrointestinal Panel — The 22-target FilmArray® GI Panel allows a syndromic approach to the diagnosis of infectious diarrhea as it includes bacteria, viruses and parasites in one test. Results are typically available within two hours of collection.

SUMMARY:
This research study will test a laboratory test called Film-Array Gastrointestinal (GI) Panel. This GI Panel is a test that can identify the bacteria or viruses that may cause diarrhea. This test will enable the ED doctor to better understand the cause of diarrhea to try to determine the best treatment.

The primary objective of this study is to determine if testing ED patients who complain of diarrhea will lead to more optimal use of antibiotics. Optimal use of antibiotics is defined as the most appropriate antibiotic to treat a specified pathogen.

ELIGIBILITY:
Inclusion Criteria:

* Presumed infectious diarrhea (3 or more loose stools in past 24 hours)
* Must have one of the 3 following features or symptoms lasting more than 7 days.

  1. Symptoms greater than 24 hours;
  2. Dehydration (defined as the need for intravenous fluid or per clinician's judgement ((based on the general appearance and alertness of the patient, the pulse, the blood pressure, the presence or absence of postural hypotension, the mucous membranes and tears, sunken eyes, skin turgor, capillary refill, and jugular venous pressure.))
  3. Inflammation (defined as fever (greater than 100.1), blood in stool per patient, DRE, or tenesmus.)

Exclusion Criteria:

* Chronic Symptoms (>14 days)
* Inability to Follow- Up (i.e. no telephone)
* Prisoner
* Likely non-infectious cause of diarrhea (Crohn's disease, radiation colitis, irritable bowel syndrome, or celiac disease)
* Confirmed C. Diff Diarrhea
* Unable to provide written consent
* Non- English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Meltzer, MD, MS, Principal Investigator — The George Washington University
Locations (1):
- The George Washington University, Department of Emergency Medicine, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Control
Started | 38 | 36
Completed | 38 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [26 to 51.25] | 33 [25.75 to 52.25] | 34 [26 to 52.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 15 | 17 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 21 | 21 | 42
  Race: White | 10 | 9 | 19
  Race: Asian, Native American, Other, Unknown | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Optimal Antibiotic Chosen
Description: Optimal use of antibiotics is defined as the most appropriate antibiotic to treat a specified pathogen. Designated physicians on study staff will retrospectively examine charts of enrolled subjects will evaluate whether the antibiotic chosen by treating clinician was appropriate given GI PCR results.
Time Frame: 30 Days post ED Discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 38 | 36
Participants | 13 | 8

2. Secondary Outcome: ED Length of Stay
Description: Time from patient arrival to time when patient is officially discharged or admitted
Time Frame: 30 Days post ED Discharge
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Experimental | Control
Number analyzed (Participants) | 38 | 36
hours | 7.68 [6.43 to 10.67] | 8.15 [5.90 to 11.23]

3. Secondary Outcome: Hospital Admission Rate
Time Frame: 30 Days post ED Discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 38 | 36
Participants | 7 | 3

4. Secondary Outcome: Rate of Abdominal/Pelvic CT Scans
Time Frame: 30 Days post ED Discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 38 | 36
Participants | 8 | 8

ADVERSE EVENTS:
Time Frame: Day 7 and Day 30
Description: No adverse events were elicited at day 7 or day 30
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/36
Other Adverse Events (participants affected / at risk) | 0/38 | 0/36

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT03809117/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT03809117/ICF_001.pdf